CLINICAL TRIAL: NCT06067282
Title: Effect of 12-week Microteaching Training on the Teaching Skills Level of University Students Majoring in Physical Education in China
Brief Title: Effect of Microteaching Training on the Teaching Skills Level of University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chai Weili (Other)
Responsible Party: Sponsor-Investigator, Chai Weili, Principal Investigator, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-K-100
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Teaching Skills
Keywords: Microteaching; Teaching Skills

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group used microteaching training to cultivate the teaching skills of university students majoring in physical education in China.
  Interventions: Other: Microteaching
- Control group (Active Comparator): The control group trained the students' teaching skills by conventional training methods.
  Interventions: Other: Microteaching

INTERVENTIONS:
Other: Microteaching — This program selects five kinds of core teaching skills for training, and the training program is extracted in "Microteaching" .

SUMMARY:
The general objective of this study is to evaluate the effect of 12-week microteaching training on the teaching skills level of university students majoring in physical education in China.

The specific objective of this study is to examine the effect of microteaching training on verbal command, movement explanation, movement demonstration, diagnostic error correction, and organization and management skills of university students majoring in physical education in China.

The participants will be divided into an experimental group and a control group. Microteaching and conventional training were used respectively to verify the influence of microteaching training on the teaching skills level of university students majoring in physical education in China.

ELIGIBILITY:
Inclusion Criteria:

1. University student
2. Major in Physical Education
3. Healthy
4. Able to perform all tests
5. Understand the study purposes and procedures
6. No previous experience performing microteaching training

Exclusion Criteria:

1. University students not majoring in Physical Education
2. Exclude participants who have not finished all tests
3. Not understanding the study purposes and procedures
4. Participants with an experience in microteaching

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Verbal command Skill Microtraining Evaluation Form | Two weeks.
  A form is used to evaluate the teacher's teaching behavior and the student's response when the teacher uses the verbal command skill.
Movement Explanation Skill Microtraining Evaluation Form | Two weeks.
  A form is used to evaluate the teacher's teaching behavior and the student's response when the teacher uses the movement explanation skill.
Movement Demonstration Skill Microtraining Evaluation Form | Two weeks.
  A form is used to evaluate the teacher's teaching behavior and the student's response when the teacher uses the movement demonstration skill.
Diagnostic error correction Skill Microtraining Evaluation Form | Two weeks.
  A form is used to evaluate the teacher's teaching behavior and the student's response when the teacher uses the diagnostic error correction skill.
Organization and Management Skill Microtraining Evaluation Form | Two weeks.
  A form is used to evaluate the teacher's teaching behavior and the student's response when the teacher uses the organization and management skill.

CONTACTS AND LOCATIONS:
Locations (1):
- Yancheng Teachers University, Yancheng, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No